CLINICAL TRIAL: NCT00526864
Title: Measuring Herpes Zoster and Post-Herpetic Neuralgia Associated Burden of Illness and Health Care Utilization and Costs in Thailand
Brief Title: Measuring Herpes Zoster and PHN Associated Burden of Illness and Health Care Utilization Costs in Thailand
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: MUTM2007-035
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Herpes Zoster
Keywords: Burden of Illness for Herpes zoster in Thailand.
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elderly patients
- HIV infected patients
- Immunosuppressed patients

SUMMARY:
Total 7 institutions will be recruited i.e. Clinical Infectious Disease Research Unit Department of Clinical Tropical Medicine, Faculty of Tropical Medicine Mahidol University,Bamrasnaradura Infectious Disease Institute

,Pramonkutklao Hospital,Rajavithi Hospital,NationalCancerInstitute,Institute of Dermatology,Raj Pracha Samasai Institute

OBJECTIVES

* Measure the burden of illness due to herpes zoster (Zoster) and post-herpetic neuralgia (PHN) (severity and duration);
* Assess the quality of life (QoL) and quality adjusted life years (QALY) lost due to Zoster and PHN;
* Describe health care resource utilization associated with Zoster and PHN;
* Describe the direct and indirect costs per case of Zoster and PHN

DETAILED DESCRIPTION:
This will be a prospective cohort study of patients presenting with Zoster rash in 7 specialized institutions in Thailand.

Subjects will be entered in the cohort at the time of presentation with Zoster rash. After the baseline assessment (day 0) that will be conducted at the investigator's office there will be 4 assessments (prospective part of the study) that will be conducted at day 7, month 1, month 3 and month 6.

We expect that there will be approximately 150 patients included in the study cohort. Cohort assembly will take place between April 2007 and October 2007.

The study will be conducted in 3 groups

Eligible patients for each group will include

* Group A: Both male and female patients ≥ 50 years of age with Zoster rash.
* Group B: Both HIV infected male and female patients ≥ 20 years of age with Zoster rash.
* Group C: Both Oncology male and female patients ≥ 20 years of age who on chemotherapy with Zoster rash.

Key exclusion criteria includes patient who refuses to sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed diagnosis of Zoster rash
* of onset of Zoster rash must be documented in the patient's chart.
* Patient is capable of understanding the study and the content of the consent form and has agreed to participate in the study by signing the informed consent.
* Patient will be available for the study follow up period

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: total of 180 clinically diagnosed herpes zoster patients, either aged ‡ 50 years and otherwise healthy, or ‡ 20 years with HIV infection, or ‡ 20 years and currently receiving chemotherapy or immunosuppressive agents.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Professor, Principal Investigator — Department of Clinical Tropical Medicine, Faculty of Tropical Medicine
Locations (1):
- Department of Clinical Tropical Medicine, Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok, Thailand